CLINICAL TRIAL: NCT05115474
Title: Phase II Study of Screening Brain MRIs in Stage IV Breast Cancer
Brief Title: Study of Screening Brain MRIs in Stage IV Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Florida Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: MCC-21448
Record Dates: First submitted 2021-11-01; First posted 2021-11-10 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Triple Negative Breast Cancer; HER2-positive Breast Cancer; Hormone Receptor-positive Breast Cancer
Keywords: Stage IV Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected to evaluate changes in surrogate biomarkers related to brain metastasis progression. Changes in biomarkers such as cytokines associated with T-cell activation and lymphocyte subpopulations may provide evidence of brain metastasis progression. Furthermore, circulating tumor DNA may identify populations of patients more likely to undergo CNS progression
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Participants with TNBC (triple negative breast cancer): Participants will undergo a screening brain MRI. Patients will undergo a second brain MRI at first systemic progression or at 6 months whichever event occurs sooner.
  Interventions: Diagnostic Test: Magnetic Resonance Imaging
- Participants with Human Epidermal Growth Factor Receptor 2 (HER2) + Breast Cancer: Participants will undergo a screening brain MRI. Patients will undergo a second brain MRI at first systemic progression or at 6 months whichever event occurs sooner.
  Interventions: Diagnostic Test: Magnetic Resonance Imaging
- Participants with Hormone Receptor (HR) +Breast Cancer: Participants will undergo a screening brain MRI. Patients will undergo a second brain MRI at first systemic progression or at 6 months whichever event occurs sooner.
  Interventions: Diagnostic Test: Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging — Participants will undergo MRI imaging with and without contrast.
  Other Names: MRI

SUMMARY:
The study is a single arm, nonrandomized phase II prospective study, with the goal of investigating the role of screening brain MRIs in neurologically asymptomatic patients with metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of breast cancer with documentation of ER/PR/HER2 status
* Radiographic evidence of stage IV extracranial diease having progressed past first line therapy in HR+/HER2- patients
* Radiographic evidence of stage IV extracranial disease in TN and HER2+ patients
* Age ≥ 18
* Life expectancy ≥ 6 months
* Eastern Cooperative Oncology Group performance status 0 to 2
* Patients must be able to understand and the willingness to sign an informed consent for study procedures
* Stated willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

* Prior diagnosis or treatment of brain metastases or leptomeningeal disease
* Patients with prior history of non-breast cancer malignancies should have no evidence of disease ≥ 2 years
* Neurologic symptoms warranting standard screening brain MRI in the judgement of the treating physician at time of enrollment
* Indications warranting brain MRI for other neurologic conditions at time of study entry
* Contraindication towards MRI imaging with contrast
* Chronic kidney disease stage IV or V or end stage renal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage IV breast cancer patients at Moffitt Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2021-12-21 (Actual); Primary Completion 2026-04-17 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Rate of Brain Metastasis | at Baseline
  Rate of brain metastasis by breast cancer subtype at baseline using MRI images.
Rate of Brain Metastasis | up to 6 months
  Rate of brain metastasis by breast cancer subtype at 6 months or first systemic progression using MRI images.

SECONDARY OUTCOMES:
Rate of Asymptomatic Leptomeningeal Disease | Baseline and at up to 6 months
  Rate of asymptomatic leptomeningeal disease by breast cancer subtype at baseline and at 6 months or first systemic progression, using MRI images.
Number of Brain Metastases | Baseline
  Number of Brain Metastases at Diagnosis by Breast Cancer Subtype, using MRI images.
Overall Survival | Up to 6 months
  Overall Survival (OS) will be measured from the initial on study date to the recorded date of death.
Number of Participants Requiring Whole Brain Radiation Therapy vs Stereotactic Radiation | Up to 6 months
  Number of Participants Requiring Whole Brain Radiation Therapy vs Stereotactic Radiation by breast cancer type.
Brain Metastasis Specific Survival | Up to 6 months
  Brain metastasis specific survival following brain metastasis by breast cancer subtype

CONTACTS AND LOCATIONS:
Overall Officials: Kamran A Ahmed, MD, Principal Investigator — Moffitt Cancer Center
Locations (2):
- United States (2):
  - Morton Plant Mease- Baycare, Clearwater, Florida
  - Moffitt Cancer Center, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ahmed KA, Kim Y, Armaghani AJ, Arrington JA, Costa RL, Czerniecki BJ, Diaz R, Dowell RA, Extermann M, Forsyth PA, Lee KT, Loftus L, Mills MN, Phuoc VH, Rosa M, Soliman HH, Sam CS, Washington IR, Soyano AE, Han HS. Phase II trial of brain MRI surveillance in stage IV breast cancer. Neuro Oncol. 2025 Jul 30;27(6):1550-1558. doi: 10.1093/neuonc/noaf018. PMID 39851040